CLINICAL TRIAL: NCT06500416
Title: Visual Outcomes Following Implantation of Tecnis Symfony Opti-Blue EDOF IOL in Patients With Mild to Moderate Retinal Ocular Comorbidities
Brief Title: Visual Outcomes of Tecnis Symfony Opti-Blue EDOF Intraocular Lens (IOL)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Coastal Eye Surgeons PLLC (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CES/OS/01/2023
Record Dates: First submitted 2024-07-09; First posted 2024-07-15 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Cataract
Keywords: Retinal comorbidity; Tecnis Symfony Optiblue Intraocular Lens
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Intervention Model Description: This prospective, non-comparative, interventional study will include 15 cataract patients (30 eyes) who will undergo femtosecond laser-assisted cataract surgery with implantation of the Tecnis Symfony OptiBlue/ Tecnis Symfony OptiBlue toric IOL in both eyes.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Tecnis Symfony OptiBlue/ Tecnis Symfony OptiBlue toric IOL (Experimental): This prospective, non-comparative, interventional study will include 15 cataract patients (30 eyes) who will undergo femtosecond laser-assisted cataract surgery with implantation of the Tecnis Symfony OptiBlue/ Tecnis Symfony OptiBlue toric IOL in both eyes.
  Interventions: Device: Tecnis Symfony OptiBlue/ Tecnis Symfony OptiBlue toric IOL

INTERVENTIONS:
Device: Tecnis Symfony OptiBlue/ Tecnis Symfony OptiBlue toric IOL — Tecnis Symfony lens (DXR00V/ZXR00V) has the OptiBlue violet light filter (VLF), which blocks short-wavelength light. Violet light filtration reduces light scatter, improving contrast and reducing nighttime visual disturbances such as halo, glare, and starbursts.

SUMMARY:
Tecnis Symfony Optiblue EDOF IOL is the latest version of Tecnis Symfony IOL with a violet light filter (VLF), which blocks short-wavelength light and improves the quality of vision while minimizing visual disturbances. The present study aims to assess the visual outcomes at distance, intermediate, and near following cataract surgery and implantation of Tecnis Symfony Optiblue IOL in patients with retinal comorbidities.

DETAILED DESCRIPTION:
Extended depth of focus (EDOF) IOLs, on the other hand, are based on the principle of creating a single-elongated focal point to enhance the depth of focus (DOF) and eliminate the overlapping of near and far images caused by traditional multifocal IOLs, thus generating a lower incidence of halos and glare. The Tecnis Symfony (Johnson & Johnson Vision) EDOF IOL incorporates a diffractive echelette design to increase the range of vision. The achromatic technology corrects chromatic aberration and increases retinal image contrast.

The latest version of the Tecnis Symfony lens (DXR00V/ZXR00V) has the OptiBlue violet light filter (VLF), which blocks short-wavelength light. Violet light filtration reduces light scatter, improving contrast and reducing nighttime visual disturbances such as halo, glare, and starbursts. As such, the present study aims to assess the visual outcomes at distance, intermediate and near following implantation of violet light filtering Tecnis Symfony Optiblue EDOF IOLs in patients with retinal comorbidities undergoing cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with retinal comorbidities, with visual acuity potential of 20/30 or better, who wish to undergo bilateral cataract surgery and are willing to provide written informed consent and adhere to study requirements.

Exclusion Criteria:

* Corneal dystrophies
* Central corneal scarring
* Keratoconus
* Proliferative diabetic retinopathy
* Exudative macular degeneration
* Zonular weakness
* Pseudoexfoliation
* Fovea-involving atrophy
* Severe dry eye
* Amblyopia
* Pupil abnormalities
* Need for an IOL outside the range of +5.0 D to +34.0 D or cylinder power over 3.75 D
* Patients who have undergone prior cataract surgery and IOL implantation in either eye; had prior corneal refractive or corneal transplantation surgery; diabetics post-vitrectomy; or who have a history of macula-off retinal detachment will also be excluded.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Binocular uncorrected visual acuity at distance | 3 months
  Mean binocular uncorrected visual acuity at distance
Binocular uncorrected visual acuity at intermediate | 3 months
  Mean binocular uncorrected visual acuity at intermediate
Binocular uncorrected visual acuity at near | 3 months
  Mean binocular uncorrected visual acuity at near

OTHER OUTCOMES:
Monocular uncorrected visual acuity at distance | 3 months
  Mean monocular uncorrected visual acuity at distance
Monocular corrected visual acuity at distance | 3 months
  Mean monocular corrected visual acuity at distance
Monocular uncorrected visual acuity at intermediate | 3 months
  Mean monocular uncorrected visual acuity at intermediate
Monocular distance-corrected visual acuity at intermediate | 3 months
  Mean monocular distance corrected visual acuity at intermediate
Monocular uncorrected visual acuity at near | 3 months
  Mean monocular uncorrected visual acuity at near
Monocular distance-corrected visual acuity at near | 3 months
  Mean monocular distance corrected visual acuity at near
Binocular corrected visual acuity at distance | 3 months
  Mean binocular corrected visual acuity at distance
Binocular distance-corrected visual acuity at intermediate | 3 months
  Mean binocular distance-corrected visual acuity at intermediate
Binocular distance-corrected visual acuity at near | 3 months
  Mean binocular distance-corrected visual acuity at near

CONTACTS AND LOCATIONS:
Locations (1):
- Coastal eye surgeons, Greenwich, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No